CLINICAL TRIAL: NCT03458819
Title: Epithelial to Mesenchymal Transition (EMT) in Peritoneal Dialysis Patients
Brief Title: EMT in Peritoneal Dialysis Patients
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 18-0401
Record Dates: First submitted 2018-02-26; First posted 2018-03-08 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Peritoneal Dialysis Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Isolated human peritoneal mesothelial cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control: Patients on neither active Vitamin D or a statin
  Interventions: Diagnostic Test: Isolation of peritoneal mesothelial cells
- Vit D: Patients on active Vitamin D but not a statin
  Interventions: Diagnostic Test: Isolation of peritoneal mesothelial cells
- Statin: Patients on a statin but not active Vitamin D
  Interventions: Diagnostic Test: Isolation of peritoneal mesothelial cells
- D + Statin: Patients on both active Vitamin D and a statin
  Interventions: Diagnostic Test: Isolation of peritoneal mesothelial cells

INTERVENTIONS:
Diagnostic Test: Isolation of peritoneal mesothelial cells — HPMCs will be isolated and stored at -80 degrees until analysis. Changes in the protein expression of EMT markers such as E-cadherin, a- SMA, Snail, and fibronectin in the HPMCs will be evaluated by Western blot analysis.

SUMMARY:
Approximately 10-11% of end stage kidney disease patients worldwide utilize peritoneal dialysis (PD) as their method of renal replacement therapy. Over time, the peritoneal membrane often undergoes anatomic and functional changes due to the process of epithelial to mesenchymal transition (EMT). EMT is characterized by increases in pro-inflammatory and pro-angiogenic cytokines. In this process, the mesothelial cells lining the peritoneal membrane are denuded and change their morphology to one more closely resembling fibroblasts. These fibroblasts invade the submesothelial zone of the peritoneal membrane resulting in marked fibrosis, and the pro-angiogenic cytokines cause an increase in neovascularization. Jointly, these processes culminate in impaired function of the peritoneal membrane and often limit the duration of effective PD therapy.

In vitro studies in cultured human peritoneal mesothelial cells (HPMCs) and in vivo studies in rodent models of PD have demonstrated that the use of active Vitamin D receptor agonists or statins may attenuate this process of EMT. These are both classes of drugs that are commonly in use by patients on PD. The investigators goal is to determine whether either or both of these drugs might attenuate the process of EMT in patients performing PD.

DETAILED DESCRIPTION:
Patients will perform a standard 2 Liter overnight dwell with the usual 2.5% dextrose PD solution. This will be done the night before a routinely scheduled visit to the home dialysis clinic. In the clinic the fluid will be drained in usual fashion and the fluid- which would otherwise be discarded- will be analyzed as below:

HPMCs will be isolated as previously described by Kinashi et al. and stored at -80 degrees until analysis. Changes in the protein expression of EMT markers such as E-cadherin, alpha smooth muscle actin (a-SMA), Snail, and fibronectin in the HPMCs will be evaluated by Western blot analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Patients on Peritoneal dialysis, and
* Patients that meet at least one of the criteria noted in the Population Description.

Exclusion Criteria:

* Patients with Recent peritonitis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PD patients > 18 years old. We propose to study 4 groups of 6 patients each:
  1. Patients taking neither an active Vitamin D analogue nor a statin
  2. Patients already taking an active Vitamin D analogue
  3. Patients already taking a statin
  4. Patients already taking both an active Vitamin D analogue and a statin
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
Changes in the protein expression of EMT markers | One year or at the end of the study, whichever occurs first.
  The goal of this study is to determine whether either or both of these drugs, Vitamin D receptor agonists or statins, might attenuate the process of EMT in peritoneal mesothelial cells. Changes in the protein expression of EMT markers such as E-cadherin, a- SMA, Snail, and fibronectin in the HPMCs will be evaluated by Western blot analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Teitelbaum, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No